CLINICAL TRIAL: NCT06149442
Title: Effectiveness of the Dry Needling Technique According to the Number of Incisions in the Treatment of Neck Pain
Brief Title: The Importance of the Number of Incisions in the Effectiveness of Dry Needling
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Principal investigator, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CEIM/2022/1/008
Record Dates: First submitted 2023-11-20; First posted 2023-11-29 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Neck Pain
Keywords: dry needling; myofascial trigger point
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose of five muscle incisions (Experimental): Subjects treated in this group will receive an in-out technique with a dosage of five incisions in the myofascial trigger point of the levator scapulae muscle.
  Interventions: Other: Dose of five-incisions dry needling technique
- Dose of ten muscle incisions (Experimental): Subjects treated in this group will receive an in-out technique with a dosage of ten incisions in the myofascial trigger point of the levator scapulae muscle.
  Interventions: Other: Dose of ten-incisions dry needling technique
- Dose of fifteen muscle incisions (Experimental): Subjects treated in this group will receive an in-out technique with a dosage of fifteen incisions in the myofascial trigger point of the levator scapulae muscle.
  Interventions: Other: Dose of fifteen-incisions dry needling technique

INTERVENTIONS:
Other: Dose of five-incisions dry needling technique — Once we have assessed the existence of a myofascial trigger point in the levator scapulae muscle, and while the subject is in lateral decubitus on the same side, with a forceps palpation, we apply a rapid in /out dry needling technique (five incisions).
  Arms: Dose of five muscle incisions
Other: Dose of ten-incisions dry needling technique — Once we have assessed the existence of a myofascial trigger point in the levator scapulae muscle, and while the subject is in lateral decubitus on the same side, with a forceps palpation, we apply a rapid in /out dry needling technique (ten incisions).
  Arms: Dose of ten muscle incisions
Other: Dose of fifteen-incisions dry needling technique — Once we have assessed the existence of a myofascial trigger point in the levator scapulae muscle, and while the subject is in lateral decubitus on the same side, with a forceps palpation, we apply a rapid in /out dry needling technique (fifteen incisions).
  Arms: Dose of fifteen muscle incisions

SUMMARY:
The dry needling technique is a procedure increasingly used by health professionals.

Dry needling consists of the use of a filiform needle to treat musculoskeletal pain. Currently, the mechanisms by which it is an effective technique are not well understood. One of the aspects not yet evaluated is the best dose in terms of the number of times it is necessary to insert the needle into the patient to achieve the best result.

This research work aims to assess which treatment obtains the best results in the management of patients with chronic neck pain.

DETAILED DESCRIPTION:
With the objective of demonstrating how the dose used during the application of the dry needling technique is related to the effectiveness of the treatment, we have designed a study where three different doses of the dry needling technique for the treatment of myofascial trigger points will be compared in the upper trapezius muscle in participants with neck pain.

Randomly, the participants will be distributed to each of the treatment groups and we will measure how the effectiveness of each of the applied doses determines the result of the application of the dry needling technique in the treatment of neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Nonspecific mechanical neck pain for more than 3 months.
* Neck pain of at least VAS 5/10.
* Reproduction of pain and symptoms subjects on palpation.
* Pain on passive stretching of the muscle.

Exclusion Criteria:

* Subjects with previous surgical intervention.
* Subjects undergoing other intervention (rehabilitation/medication).
* Positive findings that raise suspicion of cervical radiculopathy:
* Subjects diagnosed: degenerative arthropathies, inflammatory, systemic conditions (fibromyalgia).
* Cardiovascular diseases.
* Whiplash or whiplash.
* Belenophobia.
* Dizziness and vertigo.
* Pregnant.
* Thyroid disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Neck pain | Change From Baseline in Pain Scores on the Visual Analog Scale at one month.
  Visual Analog Scale (VAS). VAS is a unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between patients with similar conditions. It is a straight horizontal line of fixed length, usually 100 mm where 0 is no pain and 10 is the worst possible pain.

SECONDARY OUTCOMES:
Disability (Neck disability index) | Change From Baseline in Pain Scores on the Visual Analog Scale at one month.
  This questionnaire has been designed to give us information as to how your neck pain has affected your ability to manage in everyday life. It´s value ranges from 0 to 10 to 50 points, where 0 is the absence of disability and 50 is the highest degree of disability.
Pain catastrophizing | Change From Baseline in Pain Scores on the Visual Analog Scale at one month.
  Pain Catastrophizing Scale (PCS). The PCS is a 13-item instrumen that task participants to reflect on past painful experiences, and to indicate the degree to which they experienced each of 13 thoughts or feelings when experiencing pain, on 5-point scales with the end points (0) not at all and (4) all the time. The PCS total scores range from 0 - 52. 0 is the best result and 52 is the worst result.
kinesiophobia | Change From Baseline in Pain Scores on the Visual Analog Scale at one month.
  The Tampa Scale of Kinesiophobia (TSK) describe patient circumstances characterised by an "excessive, irrational, and debilitating fear of physical movement and activity resulting from a feeling of vulnerability to painful injury or reinjury. The TSK is a 17 item assessment checklist.The 17 item TSK total scores range from 17 to 68 where the lowest 17 means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia.
The Global Rating of Change (GRoC) | Change From Baseline in Pain Scores on the Visual Analog Scale at one month.
  It's a scale that assesses whether the patient condition has gotten worse, better, or stayed

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pecos-Martin, PhD, Study Director — Alcalá University
Locations (2):
- Spain (2):
  - Centro Investigación Fisioterapia y Dolor, Alcalá de Henares, Madrid
  - Physiotherapy and Pain Institute, Alcalá de Henares, Madrid